CLINICAL TRIAL: NCT04276961
Title: Acupuncture in Addition to Usual Care for the Treatment of Refractory Irritable Bowel Syndrome: a Randomized Controlled Trial
Brief Title: Efficacy of Acupuncture in Refractory Irritable Bowel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Collaborators: Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, zheng hui, Clinical Professor, Chengdu University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019YFC1709004
Record Dates: First submitted 2020-02-14; First posted 2020-02-19 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture plus usual care (Experimental): Acupuncture will be given on the basis of usual care. A total of 12 sessions of acupuncture will be given over a period of 4 weeks.
  Interventions: Other: Acupuncture
- Sham acupuncture plus usual care (Sham Comparator): Sham acupuncture refers to acupuncture at sham points. Sham acupuncture will be given on the basis of usual care. A total of 12 sessions of sham acupuncture will be given over a period of 4 weeks.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Acupuncture will be given for a total of 12 session over 4 weeks. Acupuncture at acupoints Tianshu (ST25), Shangjuxu (ST37), Zusanli (ST36), and Neiguan (PC6) bilaterally will be given.

SUMMARY:
The trial aims to examine the efficacy and safety of acupuncture in the treatment of refractory irritable bowel syndrome (IBS). The investigators will include 170 participants to receive acupuncture plus usual care or sham acupuncture plus usual care. Twelve sessions of acupuncture will be delivered to participants over a period of 4 weeks. The primary outcome is defined as proportion of participants with adequate relief of global IBS symptoms at week 8, which is defined as >50% reduction in IBS-SSS scale.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-70 years (either sex);
* Fulfilled Rome IV criteria for IBS;
* Patients with normal occult blood in stool in recent one month;
* The age is above 50, the results of colonoscopy are normal in near year;
* Symptoms are present for ≥12 months;
* There is an absence of response to a minimum of 6 weeks of dietary intervention or advice;
* There is an absence of response to an adequate dose of at least one conventional pharmacological agent tried for a minimum of 6 weeks;
* Signed the written informed consent form.

Exclusion Criteria:

* Previous colonoscopy, meal barium fluoroscopy, abdominal ultrasound and other examinations found severe intestinal organic lesions (including but not limited to ulcerative colitis, familial multiple intestinal polyps, colorectal cancer patients);
* The presence of one or more of the following warning symptoms: unexplained rectal bleeding, a positive faecal occult blood test result; anaemia, abdominal mass, ascites, fever, and emaciation;
* The presence of other severe medical conditions, such as cardiovascular disease, endocrine disorders, hepatic dysfunction, renal diseases, and cognitive disorders that can affect the outcome assessment results;
* Unconscious, unable to express subjective symptoms of discomfort and clearly diagnosed severe mental disorders;
* An unstable psychological state or accompanying psychological disorders (SDS>56);
* With pregnancy or lactation;
* Accepting acupuncture treatment in the last 3 months;
* Difficulties in attending the trial, such as fear of acupuncture.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants with adequate relief of global IBS symptoms | 4 weeks after randomization (week 4)
  Adequate relief of global IBS symptoms will be defined as a >50% reduction in the IBS symptom severity scale (IBS-SSS).

SECONDARY OUTCOMES:
IBS symptom severity scale | Baseline (week 0), week 2, 4, 6, 8
  The IBS symptom severity scale (IBS-SSS) has a total of 500 points. The score ranges from 0 to 500; higher scores indicating more severe symptoms; a score over 300 indicates severe symptoms.
Weekly bowel movements | Baseline (week 0), week 2, 4, 6, 8
  The total number of bowel movements in a week.
Work and Social Adjustment Scale | Baseline (week 0), week 2, 4, 6, 8
  The Work and Social Adjustment Scale (WSAS) measures the effect of IBS on ability to work and manage at home, participate in social and private leisure activities and maintain relationships. It has five domains scored 0 (not affected) to 8 (severely affected), with a total possible score of 40.
Irritable Bowel Syndrome Quality of Life Instrument | Baseline (week 0), week12, and month12
  Irritable Bowel Syndrome Quality of Life Instrument (IBS-QOL) is a condition-specific measure for assessing health-related QoL among persons with irritable bowel syndrome. The IBS-QOL had eight subscales. The IBS-QOL and its subscales were both scored on a range of 0-100 with higher scores suggestive of better QOL.
Bristol Stool Form Scale | Baseline, weeks 2, 4, 6 and 8.
  The Bristol Stool Form Scale is a tool that is used for the assessment of stool consistency. Scores 1-2 indicate constipation, scores 3-5 indicate normal stool; scores 6-7 indicate diarrhea.
Self-Rating Anxiety Scale (SAS) | Baseline, weeks 2, 4.
  The SAS is a self rating scale for the assessment of the severity of anxiety.
Self-Rating Depression Scale (SDS) | Baseline, weeks 2, 4.
  The SDS is a self rating scale for the assessment of the severity of depression.

OTHER OUTCOMES:
Proportion of participants with adverse events | Week 4 and 12
  Side effect of acupuncture or sham acupuncture will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Gang Li, MD, Principal Investigator — Beijing University of Chinese Medicine
Locations (1):
- Hospital of Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Conditional share, the principle investigator will ask for the reasons to use the data.
Supporting Information: Study Protocol
Time Frame: After the completing the study for 2 years

REFERENCES:
- [Derived] Zhao J, Chen M, Wang X, Ye K, Shi S, Li H, Wang J, Chen X, Ni J, Wei Q, Shi Y, Hu Y, Sun J, Li D, Liu S, Li Z, Zheng H, Yu SG. Efficacy of acupuncture in refractory irritable bowel syndrome: study protocol for a randomised controlled trial. BMJ Open. 2021 Sep 13;11(9):e045655. doi: 10.1136/bmjopen-2020-045655. PMID 34518248